CLINICAL TRIAL: NCT00608023
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled Extension Study Assessing the Efficacy and Long-term Safety of a 2 mg Dose of TH9507, a GHRH Analog, in HIV Subjects With Excess Abdominal Fat Accumulation
Brief Title: TH9507 Extension Study in Patients With HIV-Associated Lipodystrophy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Theratechnologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TH9507-CTR-1012
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Results first posted 2014-01-15 (Estimated); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Lipodystrophy; HIV Infections
Keywords: HIV; Lipodystrophy; Abdominal fat accumulation; Growth hormone releasing hormone; HIV-associated lipodystrophy; Treatment experienced
MeSH Terms: conditions — Lipodystrophy; HIV Infections; HIV-Associated Lipodystrophy Syndrome | interventions — tesamorelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Tesamorelin 12 months (T-T) (Experimental): Tesamorelin 2 mg/day for 12 months
  Interventions: Drug: Tesamorelin
- Tesamorelin-Placebo (T-P) (Experimental): Tesamorelin 2 mg/day for 6 months - Placebo for 6 months
  Interventions: Drug: Tesamorelin; Drug: Placebo for Tesamorelin
- Placebo-Tesamorelin (P-T) (Experimental): Placebo 6 months - Tesamorelin 2 mg/day for 6 months
  Interventions: Drug: Tesamorelin; Drug: Placebo for Tesamorelin

INTERVENTIONS:
Drug: Tesamorelin
  Other Names: Egrifta
Drug: Placebo for Tesamorelin
  Arms: Placebo-Tesamorelin (P-T); Tesamorelin-Placebo (T-P)

SUMMARY:
Assessing the Efficacy and Long-Term Safety of a 2 mg dose of TH9507, a Growth Hormone-Releasing Factor Analog, in HIV Subjects with Excess Abdominal Fat Accumulation

DETAILED DESCRIPTION:
HIV lipodystrophy affects a significant proportion of patients treated with combination antiretroviral therapy (ART) and is characterized by excess visceral fat accumulation, loss of extremity and subcutaneous fat, in association with dyslipidemia and insulin resistance. Data from the first Phase 3 multicenter, randomized, placebo-controlled trial demonstrated that daily administration of 2mg TH9507, a growth hormone releasing factor (GRF), to HIV- infected patients with excess of abdominal fat accumulation for 26 weeks resulted in decreases in visceral adipose tissue (VAT) and trunk fat, with lesser changes in limb fat and subcutaneous adipose tissue (SAT). The present study is aimed at confirming the observations made during the first Phase 3 study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have completed the 26 weeks treatment period of the TH9507-CTR-1011 study.
* Signed informed consent before any trial-related activities.

Exclusion Criteria:

* Fasting blood glucose >8.33 mmoL (150 mg/dL) at the end of the TH9507-CTR-1011 study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2007-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Grinspoon, MD, Principal Investigator — Massachusetts General Hospital
Locations (47):
- United States (27):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Body Positive Inc., Phoenix, Arizona
  - Somero, Michael, Indio, California
  - UCLA School of Medicine, Los Angeles, California
  - Office of Dr. Michael Somero, Palm Springs, California
  - University of California, San Francisco, California
  - Kaiser Permanente, San Francisco, California
  - UCSF/VA Medical Center, San Francisco, California
  - AIDS Research Alliance, West Hollywood, California
  - Denver Public Health Department, Denver, Colorado
  - Office of Dr. Gary Richmond, Fort Lauderdale, Florida
  - Hendry/Glades County Health Departments, LaBelle, Florida
  - Infectious Disease Research Institute Inc., Tampa, Florida
  - AIDS Research Consortium Atlanta (ARCA), Atlanta, Georgia
  - Northern Healthcare, Chicago, Illinois
  - Northstar Medical, Chicago, Illinois
  - Indiana University Department of Medicine, Indianapolis, Indiana
  - Tufts University School of Medicine, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - The Research Institute, Springfield, Massachusetts
  - ID Associates, Hillsborough, New Jersey
  - AIDS Community Research Initiative of America, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Central Texas Clinical Research, Austin, Texas
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Swedish Medical Center, Seattle, Washington
- C. H. U. Sart-Tilman, Liège, Belgium
- Canada (7):
  - St-Paul's Hospital, Vancouver, British Columbia
  - McMaster University Health Sciences Centre, Hamilton, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Centre Hospitalier Universitaire de Santé de l'Estrie, Fleurimont, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Groupe de Recherche en Rhumatologie et maladies osseuses, Ste-Foy, Quebec
- France (4):
  - Hôpital Hotel Dieu Lyon, Lyon
  - Hotel Dieu, Nantes
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Necker, Paris
- Spain (3):
  - Hosp. Ramon y Cajal, Madrid
  - Hosp. Clinico San Carlos, Madrid
  - Hosp.C.U.de Santiago, Santiago de Compostela
- United Kingdom (5):
  - BSUH NHS Trust, Brighton
  - St Georges Hospital, London
  - Royal Free Hospital, London
  - Chelsea and Westminster Hospital, London
  - St Mary's NHS Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fourman LT, Czerwonka N, Feldpausch MN, Weiss J, Mamputu JC, Falutz J, Morin J, Marsolais C, Stanley TL, Grinspoon SK. Visceral fat reduction with tesamorelin is associated with improved liver enzymes in HIV. AIDS. 2017 Oct 23;31(16):2253-2259. doi: 10.1097/QAD.0000000000001614. PMID 28832410
- [Derived] Stanley TL, Falutz J, Marsolais C, Morin J, Soulban G, Mamputu JC, Assaad H, Turner R, Grinspoon SK. Reduction in visceral adiposity is associated with an improved metabolic profile in HIV-infected patients receiving tesamorelin. Clin Infect Dis. 2012 Jun;54(11):1642-51. doi: 10.1093/cid/cis251. Epub 2012 Apr 10. PMID 22495074
- [Derived] Falutz J, Mamputu JC, Potvin D, Moyle G, Soulban G, Loughrey H, Marsolais C, Turner R, Grinspoon S. Effects of tesamorelin (TH9507), a growth hormone-releasing factor analog, in human immunodeficiency virus-infected patients with excess abdominal fat: a pooled analysis of two multicenter, double-blind placebo-controlled phase 3 trials with safety extension data. J Clin Endocrinol Metab. 2010 Sep;95(9):4291-304. doi: 10.1210/jc.2010-0490. Epub 2010 Jun 16. PMID 20554713
- [Derived] Falutz J, Potvin D, Mamputu JC, Assaad H, Zoltowska M, Michaud SE, Berger D, Somero M, Moyle G, Brown S, Martorell C, Turner R, Grinspoon S. Effects of tesamorelin, a growth hormone-releasing factor, in HIV-infected patients with abdominal fat accumulation: a randomized placebo-controlled trial with a safety extension. J Acquir Immune Defic Syndr. 2010 Mar;53(3):311-22. doi: 10.1097/QAI.0b013e3181cbdaff. PMID 20101189

RESULTS

PARTICIPANT FLOW:
Groups:
- Tesamorelin (52 Weeks): Tesamorelin 2 mg/day for 52 Weeks
- Tesamorelin (26 Weeks) - Placebo (26 Weeks): Tesamorelin 2 mg/day for 26 weeks followed by Placebo for 26 weeks
- Placebo-Tesamorelin (P-T): Placebo for 26 weeks followed by Tesamorelin 2 mg/day for 26 weeks
Period: Overall Study
Arm/Group | Tesamorelin (52 Weeks) | Tesamorelin (26 Weeks) - Placebo (26 Weeks) | Placebo-Tesamorelin (P-T)
Started | 92 | 85 | 86
Completed | 80 | 63 | 72
Not Completed | 12 | 22 | 14
Not completed — Withdrawal by Subject | 8 | 10 | 7
Not completed — Adverse Event | 1 | 4 | 5
Not completed — Lost to Follow-up | 2 | 2 | 1
Not completed — Protocol Violation | 1 | 3 | 1
Not completed — Unknown reason | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Tesamorelin 52 Weeks: Tesamorelin 2 mg/day for 52 weeks
- Placebo (26 Weeks) - Tesamorelin (26 Weeks): Placebo for 26 weeks followed by Tesamorelin 2 mg/day for 26 weeks
- Total: Total of all reporting groups
Arm/Group | Tesamorelin 52 Weeks | Tesamorelin (26 Weeks) - Placebo (26 Weeks) | Placebo (26 Weeks) - Tesamorelin (26 Weeks) | Total
Number analyzed (Participants) | 92 | 85 | 86 | 263
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (6.9) | 48.9 (7.2) | 48.4 (7.9) | 48.3 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 11 | 29
  Male | 83 | 76 | 75 | 234

OUTCOME MEASURES:

1. Secondary Outcome: Changes From Baseline in Visceral Adipose Tissue (VAT) at Week 52
Description: Visceral adipose tissue (VAT) was assessed by computerized tomography (CT) scan using a single-slice. Changes in VAT between baseline and Week 52 are reported.
Time Frame: Baseline and Week 52
Population: All data were included in the analysis by intention to treat principles. Intent to treat populations were defined as all randomized subjects who were exposed to study drug (i.e injection of at least 1 dose of study drug).
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Tesamorelin 52 Weeks | Tesamorelin (26 Weeks) - Placebo (26 Weeks) | Placebo (26 Weeks) - Tesamorelin (26 Weeks)
Number analyzed (Participants) | 92 | 85 | 86
cm^2 | -41 (57) | 0 (53) | -26 (47)
Statistical Analysis 1: Comparison: Tesamorelin 52 Weeks vs Tesamorelin (26 Weeks) - Placebo (26 Weeks); Test type: Superiority or Other; p < 0.001, ANCOVA

2. Other Pre Specified Outcome: Changes From Baseline in Triglycerides at Week 52
Description: Blood lipid levels were determined under fasting conditions. Changes in triglycerides between baseline and Week 52 are reported.
Time Frame: Baseline and Week 52
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tesamorelin (52 Weeks) | Tesamorelin (26 Weeks) - Placebo (26 Weeks) | Placebo (26 Weeks) - Tesamorelin (26 Weeks)
Number analyzed (Participants) | 92 | 85 | 86
mg/dL | -37 (196) | 4 (177) | 1 (120)
Statistical Analysis 1: Comparison: Tesamorelin (52 Weeks) vs Tesamorelin (26 Weeks) - Placebo (26 Weeks); Test type: Superiority or Other; p > 0.05, ANCOVA

3. Other Pre Specified Outcome: Changes From Baseline in Total Cholesterol/HDL Cholesterol Ratio at Week 52
Description: Blood lipid levels were determined under fasting conditions. Total Cholesterol/HDL Cholesterol Ratio was obtained by dividing the total cholesterol value by the value of the HDL cholesterol. Changes between baseline and Week 52 are reported.
Time Frame: Baseline and Week 52
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Tesamorelin 52 Weeks | Tesamorelin (26 Weeks) - Placebo (26 Weeks) | Placebo (26 Weeks) - Tesamorelin (26 Weeks)
Number analyzed (Participants) | 92 | 85 | 86
ratio | -0.23 (1.75) | 0.13 (1.19) | 0.06 (1.01)
Statistical Analysis 1: Comparison: Tesamorelin 52 Weeks vs Tesamorelin (26 Weeks) - Placebo (26 Weeks); Test type: Superiority or Other; p > 0.05, ANCOVA

4. Primary Outcome: Changes From Baseline in Fasting Blood Glucose at Week 52
Description: Blood glucose was determined after an overnight fast. Changes in blood glucose between baseline and Week 52 are reported.
Time Frame: Baseline and Week 52
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tesamorelin 52 Weeks | Tesamorelin (26 Weeks) - Placebo (26 Weeks) | Placebo (26 Weeks) - Tesamorelin (26 Weeks)
Number analyzed (Participants) | 92 | 85 | 86
mg/dL | 0 (16) | -2 (34) | 1 (21)
Statistical Analysis 1: Comparison: Tesamorelin 52 Weeks vs Tesamorelin (26 Weeks) - Placebo (26 Weeks); Test type: Superiority or Other; p > 0.05, ANCOVA

5. Primary Outcome: Changes From Baseline in 2 h Oral Glucose Tolerance Test (OGTT) at Week 52
Description: Glucose tolerance was determined after an overnight fast using standard 75 gram-oral glucose tolerance test (OGTT) with glucose measured at timepoints 0, 30, 60, 90 and 120. Changes in glucose tolerance between baseline and Week 52 are reported.
Time Frame: Baseline and Week 52
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tesamorelin 52 Weeks | Tesamorelin (26 Weeks) - Placebo (26 Weeks) | Placebo (26 Weeks) - Tesamorelin (26 Weeks)
Number analyzed (Participants) | 92 | 85 | 86
mg/dL | -2 (38) | 2 (35) | 7 (37)
Statistical Analysis 1: Comparison: Tesamorelin 52 Weeks vs Tesamorelin (26 Weeks) - Placebo (26 Weeks); Test type: Superiority or Other; p > 0.05, ANCOVA

ADVERSE EVENTS:
Arm/Group | Tesamorelin 52 Weeks | Tesamorelin (26 Weeks) - Placebo (26 Weeks) | Placebo (26 Weeks) - Tesamorelin (26 Weeks)
Serious Adverse Events (participants affected / at risk) | 3/92 | 1/85 | 3/86
Other Adverse Events (participants affected / at risk) | 17/92 | 11/85 | 28/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tesamorelin 52 Weeks (N=92) | Tesamorelin (26 Weeks) - Placebo (26 Weeks) (N=85) | Placebo (26 Weeks) - Tesamorelin (26 Weeks) (N=86)
Retinopathy (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0
Hodgkin disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tesamorelin 52 Weeks (N=92) | Tesamorelin (26 Weeks) - Placebo (26 Weeks) (N=85) | Placebo (26 Weeks) - Tesamorelin (26 Weeks) (N=86)
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 5
Injection site erythema (General disorders) | 3 | 0 | 5
Injection site pain (General disorders) | 0 | 0 | 5
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 3
Musculosketal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 5
Paresthesia (Nervous system disorders) | 2 | 3 | 5
Insomnia (Psychiatric disorders) | 0 | 0 | 5

LIMITATIONS AND CAVEATS:
As this trial was completed in October 2008 hence, the primary Completion Date is prior to January 18, 2017, therefore the Protocol, and Statistical Analysis Plan have not been uploaded to the Document Section.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less